CLINICAL TRIAL: NCT05419167
Title: STEP-COVID: A Program for Pregnant Women During the SARS-CoV-2 Pandemic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government)
Responsible Party: Principal Investigator, Nicolas Berthelot, Full professor, Université du Québec à Trois-Rivières
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STEP COVID
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Psychological; Mental Health Issue; Prenatal Stress; Maternal Distress; COVID-19 Pandemic
Keywords: Mentalization; Well-being; Pregnancy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP-COVID (Experimental): Participants will participate online to the 6 sessions of the program addressing the psychological experience of pregnancy and supporting reflective capacities.
  Interventions: Behavioral: STEP-COVID
- Usual prenatal cares (No Intervention): Participants of the comparison group will receive usual prenatal cares (ex. prenatal classes)

INTERVENTIONS:
Behavioral: STEP-COVID — The program is offered by two facilitators to groups of three to six women, online in a synchronous mode. The intervention is divided into two phases, each including three sessions. The first 3 sessions aim to explore how the participants feel, to better understand what makes them feel this way, to allow them to exchange with other people who are going through similar experiences, and to support the ability to manage stress and more unpleasant emotions. The following three sessions aim to enable participants to refocus on their experience of pregnancy and motherhood by giving them the opportunity to reflect upon how they wish to be as mothers, upon how their personal history influences their experience of pregnancy and motherhood, upon the moments that, as mothers, might be the most pleasant and those that will require more adaptations, and upon identifying the needs they have or expect to have after childbirth as well as the resources available to them to meet these needs.
  Arms: STEP-COVID

SUMMARY:
STEP-COVID (Supporting the Transition to and Engagement in Parenthood during the COVID-19 pandemic) is a manualized group intervention for pregnant women during the COVID-19 pandemic designed to foster emotion regulation and reflective capacities in participants.

DETAILED DESCRIPTION:
The program aims to (a) support mentalization in relation to oneself, motherhood and the relationship with the child to be born, (b) reduce isolation by allowing participants to exchange about the positive aspects and the challenges of pregnancy and motherhood with other women, (c) explore what pregnant women are going through in the context of the pandemic, (d) allow participants to repossess their experience of pregnancy in the current context of insecurity and fear, and (e) consider new ways of coping with stress and unpleasant emotions. The program is manualized and uses structured activities based on theoretical grounds and empirical research during which facilitators share information, animate reflective activities, and facilitate exchanges.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18+ years
* Interested in reflecting about their experience of pregnancy and willing to attend weekly sessions in group setting.
* Must speak French as their first language

Exclusion Criteria:

* Severe psychiatric disorders (schizophrenia, bipolar disorder)
* Severe emotional dysregulation
* Current self-harm
* Not sure to keep the child
* High level of hostility

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change in psychological distress from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire (Kessler Distress Scale) assessing psychological distress. Change between baseline and end of pregnancy will be assessed, as well as between baseline and 6-month postpartum.
Perception of change in domains of functioning during pregnancy | Administered at one time-point, at the end of the third trimester of pregnancy. The participant will report on perceived changes during the last 9 months.
  We developed an instrument assessing one's perception of change (negative change to positive change) across multiple domains of functioning including the quality of the relationship with the partner; the quality of the relationship with significant others, self-esteem; emotion recognition, regulation and expression; social support and parental confidence. These domains will be assessed separately.
Post-traumatic growth | Administered at one time-point, at the end of the third trimester of pregnancy. The measure will assess current level of post-traumatic growth.
  Participants are invited to complete a self-report questionnaire of post-traumatic growth (Post-traumatic Growth Inventory) at the end of the third trimester of pregnancy. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Level of satisfaction concerning the intervention | Satisfaction assessed after each session of the program and after its ending. Satisfaction is thus assessed between the second trimester of pregnancy and 36-weeks of pregnancy, for a total time frame up to 7-months.
  Participants are invited to complete a self-report questionnaire assessing their level of satisfaction after each session and at the end of the program, using a Likert scale. A semi-structured interview is also administered at the end of the program that will provide qualitative information regarding their appreciation of the program.
Change in affective states from baseline (2nd trimester of pregnancy) to the end of the third trimester of pregnancy (around 36 weeks) and from baseline to 6-months postpartum | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  Participants are invited to complete a self-report questionnaire (Positive and Negative Affect Scale) assessing positive and negative affects. Change between baseline and end of pregnancy will be assessed as well as between baseline and 6-month postpartum.

SECONDARY OUTCOMES:
Parental reflective functioning | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of reflective functions.
  Participants will complete the Parental Reflective Functioning Questionnaire (PRFQ) at 6 months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Change in reflective functioning | Data will be collected at recruitment (2nd trimester of pregnancy), at 36-weeks of pregnancy and at 6-months postnatal. The assessment time frame thus covers a period of 13 months.
  The Reflective Functioning Questionnaire (RFQ-8) will be administered at baseline, at the end of the third trimester of pregnancy and at 6-months postpartum. Change between time-points will be assessed.
Change in perception of parental competence | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. The assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of maternal confidence (Maternal confidence questionnaire). Change between baseline and the end of pregnancy will be assessed.
Change in antenatal attachment | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. The assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of antenatal attachment (Maternal antenatal attachment scale). Change between baseline and the end of pregnancy will be assessed.
Self-compassion | Administered at one time-point, at the end of the third trimester of pregnancy. The measure will assess current level of self-compassion.
  Participants are invited to complete a self-report questionnaire of self-compassion (Self-Compassion Scale) at the end of the third trimester of pregnancy. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Connection to care | From the third trimester of pregnancy to 6 months postpartum. The assessment time frame thus covers a period of 7 months.
  Participants will be referred to community agencies for resources based on need during their participation to STEP. Their utilization of other resources will be assessed using self-reported questionnaires at the end of the third trimester of pregnancy and at 6 months postpartum.
Change in emotion regulation strategies | Data will be collected at recruitment (2nd trimester of pregnancy) and at 36-weeks of pregnancy. he assessment time frame thus covers a period of 7 months.
  Participants are invited to complete a self-report questionnaire of emotion regulation strategies (Cognitive Emotion Regulation Questionnaire). Change between baseline and the end of pregnancy, as well as between baseline and 6 months postpartum will be assessed.
Parental stress | Administered at one time-point, at the 6-months postpartum assessment. The measure will assess current level of parental stress.
  Participants are invited to complete a self-report questionnaire of parental stress (Parenting Stress Index) at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Maternal bonding | Administered at one time-point, at the 6-months postpartum assessment. The measure will assess current level of maternal bonding.
  Participants are invited to complete a self-report questionnaire of maternal bonding (Maternal postnatal attachment scale) at 6-months postpartum. Scores in participants to the intervention will be compared to scores of matched controls who did not participate to the intervention.
Infant general development | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of infant development.
  The Age and Stage Questionnaire Third Edition (ASQ-3) will be administered at 6-months postnatal to assess infant development.
Infant socio-emotional development | Administered at one time-point, at 6-moths postpartum. The measure will assess current level of infant development.
  The Ages & Stages Questionnaires: Social-Emotional, Second Edition (ASQ:SE-2) will be administered at 6-months postnatal to assess infant socio-emotional development.
Infant temperament | Administered at one time-point, at 6-moths postpartum.The measure will assess current infant temperament
  The Infant Behavior Questionnaire (IBQ) will be administered at 6-months postnatal to assess infant temperament

OTHER OUTCOMES:
Personality dysfunctions | Administered at one time-point, at the second trimester of pregnancy. The measure will assess current level of personality dysfunctions.
  Personality dysfunctions are assessed at baseline and will be considered as a moderator of the intervention effectiveness. Personality dysfunctions will be measured using the Self and Interpersonal Functioning Rating Scale, a 24-item self-report questionnaire designed to assess the four core elements of personality pathology (Identity, Self-direction, Empathy, and Intimacy) from the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Level of Personality Functioning for personality disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berthelot N, Garon-Bissonnette J, Drouin-Maziade C, Bergeron V, Series T. STEP-COVID: a pilot study of a prenatal intervention for pregnant women during the COVID-19 pandemic. Sci Rep. 2023 Apr 20;13(1):6466. doi: 10.1038/s41598-023-33369-8. PMID 37081093